CLINICAL TRIAL: NCT06748378
Title: Analysis of Gait Parameters After Therapy Using the Tilt-table Exercise and Motor Imagery - a Randomized Observational Study on Stroke Patients.
Brief Title: Gait Parameters After Using the Tilt-table Exercise and Motor Imagery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Olczak (Other)
Responsible Party: Sponsor-Investigator, Anna Olczak, PhD; Senior Specjalist of the Rehabilitation Clinic, Military Institute od Medicine National Research Institute
Organization: Military Institute od Medicine National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/KRN/2020
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Visualization; Gait Analysis
Keywords: gait analysis; Erigo Pro; motor imagery; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Allocation Randomized Interventional Model Parallel Assignment Masking Double (Participant Outcomes Assessor) Primary Purpose Treatment
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional rehabilitation (Experimental): In conventional rehabilitation, patients performed daily physiotherapy, which included intensive preparatory training for standing and sitting positions, strengthening exercises, weight-bearing exercises, and balance and coordination exercises (from 40 to 60 minutes of therapy).
  Interventions:
  Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery
  Interventions: Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery on gait.; Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery on gait parameters.
- Erigo®Pro (Experimental): Interventions: Effective therapy included 1 session on a tilting table at an angle of 42° for 20 minutes, 5 times a week (Monday to Friday) at a speed of 32 steps per minute, followed by a physiotherapy session for two weeks.
  Interventions:
  Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery
  Interventions: Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery on gait.; Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery on gait parameters.
- motor imagery (MI) (Experimental): in addition to conventional physiotherapy, activity imagery during passive walking on the Erigo®Pro table was introduced. During the exercises on the table, the patients wore headphones that blocked out any external sounds, closed their eyes and their task was to imagine the sensation of their body moving (first-person imagination), differentiating the idea of walking in various real environments (park, forest, beach, snow, streets). in the city, walking at different speeds, going up and down stairs, running, etc.).
  Interventions:
  Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery
  Interventions: Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery on gait.; Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery on gait parameters.

INTERVENTIONS:
Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery on gait. — 66 stroke patients were randomly assigned to three groups (22 people each) with different therapies (conventional, with the addition of Erigo®Pro and enriched with motor imagery). The therapy duration was two weeks. Patients underwent assessment before and after completion of therapy. The study used the Trunk Stability Test, and the Riablo device to measure gate parameters. Additionally, an evaluation of the superficial tension of the transverse abdominis and multifidus muscles was conducted.
Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery on gait parameters. — 66 stroke patients were randomly assigned to three groups (22 people each) with different therapies (conventional, with the addition of Erigo®Pro and enriched with motor imagery). The therapy duration was two weeks. Patients underwent assessment before and after completion of therapy. The study used the Trunk Stability Test, and the Riablo device to measure the gate parameters. Additionally, an evaluation of the superficial tension of the transverse abdominis and multifidus muscles was conducted.

SUMMARY:
Sixty-six stroke patients were randomly assigned to three groups (conventional, with the addition of the Erigo®Pro table, and enriched with motor imagery). The Trunk Stability Test, walking speed, step symmetry, and lower limb load symmetry on the Riablo device, as well as the superficial tension of the transverse abdominis and multifidus muscles, were assessed before and after completing therapy.

DETAILED DESCRIPTION:
Sixty-six stroke patients were randomly assigned to three groups (conventional, with the addition of the Erigo®Pro table, and enriched with motor imagery). The Trunk Stability Test, walking speed, step symmetry, and lower limb load symmetry on the Riablo device, as well as the superficial tension of the transverse abdominis and multifidus muscles, were assessed before and after completing therapy.

Results: In each of the groups studied, the therapies used significantly improved the functional assessment of trunk stability (Trunk Control Test <0.001)). Additionally, after the intervention, the Erigo group showed a greater gait speed (p=0.003), while the Visualization group exhibited a higher level of tension in the multifidus (p=0.011) and transverse abdominal muscles (p=0.002).

ELIGIBILITY:
Inclusion Criteria:

* 1) patients 6-8 weeks post-stroke,
* 2) aged 38-85 years, mean,
* 3) males and females,
* 4) walking with or without assistance (modified Rankin scale = 3),
* 5) with slight neurological deficits (NIHSS ≤7).

Exclusion Criteria:

* 1) stroke up to six weeks after the episode,
* 2) epilepsy,
* 3) no possibility to sit and stand,
* 4) persistent deficit of speech and cognitive functions, lack of attention,
* 5) visual disturbances,
* 6) depression,
* 7) high or very low blood pressure, dizziness, malaise.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Trunk Control Test | two weeks
  Assessment of trunk stability before and after therapy

SECONDARY OUTCOMES:
RiabloTM device | two weeks
  Assessment of gate parameters before and after therapy
Luna EMG | two weeks
  Assessment of the surface tension of the transverse abdominis muscle and the tension of the multifidus muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Military Institute of Medicine National Research Institute, Warsaw, Masovian District, Poland

IPD SHARING:
Plan to Share IPD: Undecided